CLINICAL TRIAL: NCT03846583
Title: Phase Ib Trial of Tucatinib in Combination With Abemaciclib and Trastuzumab for Patients With HER2-Positive Metastatic Breast Cancer
Brief Title: Tucatinib + Abemaciclib + Herceptin for HER2+ MBC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jose Pablo Leone, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-621
Record Dates: First submitted 2019-02-13; First posted 2019-02-19 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; abemaciclib; Trastuzumab; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): * Tucatinib is administered orally twice daily
  * Abemaciclib is administered orally twice daily
  * Trastuzumab is adminidtered intravenously once every three weeks
  * Aromatase Inhibitor is administered orally once daily
  Interventions: Drug: Tucatinib; Drug: Abemaciclib; Drug: Trastuzumab; Drug: Aromatase Inhibitor
- Arm A: Active Brain Metastases (Experimental): * Tucatinib is administered orally twice daily
  * Abemaciclib is administered orally twice daily
  * Trastuzumab is adminidtered intravenously once every three weeks
  * Aromatase Inhibitor is administered orally once daily
  Interventions: Drug: Tucatinib; Drug: Abemaciclib; Drug: Trastuzumab; Drug: Aromatase Inhibitor
- Arm B: Surgical Resection Needed (Experimental): * Tucatinib is administered orally twice daily
  * Abemaciclib is administered orally twice daily
  * Trastuzumab is adminidtered intravenously once every three weeks
  * Aromatase Inhibitor is administered orally once daily
  Interventions: Drug: Tucatinib; Drug: Abemaciclib; Drug: Trastuzumab; Drug: Aromatase Inhibitor
- Arm C: Progressive Extracranial Disease (Experimental): * Tucatinib is administered orally twice daily
  * Abemaciclib is administered orally twice daily
  * Trastuzumab is adminidtered intravenously once every three weeks
  * Aromatase Inhibitor is administered orally once daily
  Interventions: Drug: Tucatinib; Drug: Abemaciclib; Drug: Trastuzumab; Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Tucatinib — Tucatinib is a drug that inhibits human epidermal growth factor receptor 2 (HER-2) protein, which is a protein expressed in the cancer cells. By inhibiting this protein, tucatinib may help stop or reduce the growth of the tumor
Drug: Abemaciclib — Abemaciclib is a cyclin-dependent kinase (CDK) inhibitor. CDK inhibitors work to stop cell growth.
  Other Names: Verzenio
Drug: Trastuzumab — • Trastuzumab is called a "targeted therapy" because it works by attaching itself to specific receptors on the surface of breast cancer cells, known as HER2 receptors. When Trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the immune system.
  Other Names: Herceptin
Drug: Aromatase Inhibitor — These drugs act by lowering the amount of estrogen produced by the body by blocking an enzyme called aromatase

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for HER2-Postive Metastatic Breast Cancer.

The interventions involved in this study are:

* Tucatinib
* Abemaciclib (VerzenioTM)
* Trastuzumab (Herceptin®)
* Endocrine Therapy: Exemestane (Aromasin®), Letrozole (Femara®), or Anastrozole (Arimidex®)

DETAILED DESCRIPTION:
This research study is a Phase Ib clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied. The U.S. Food and Drug Administration (FDA) has not approved the combination of Tucatinib, Abemaciclib, and Trastuzumab as a treatment for any disease.

In this research study, the investigators are:

* Studying the combination of Tucatinib, Abemaciclib, Trastuzumab, and hormonal therapy.
* Tucatinib is a drug that inhibits human epidermal growth factor receptor 2 (HER-2) protein, which is a protein expressed in the cancer cells. By inhibiting this protein, tucatinib may help stop or reduce the growth of the tumor. The U.S. Food and Drug Administration (FDA) has not approved Tucatinib as a treatment for any disease, but it has been used in a research setting with humans for many years.
* Abemaciclib is a cyclin-dependent kinase (CDK) inhibitor. CDK inhibitors work to stop cell growth. The FDA has not approved Abemaciclib for this specific disease, but it has been approved for other uses.
* Trastuzumab is called a "targeted therapy" because it works by attaching itself to specific receptors on the surface of breast cancer cells, known as HER2 receptors. When Trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by your immune system. This process allows trastuzumab to help slow or stop the growth of the breast cancer. The FDA has approved Trastuzumab as a treatment for this disease.
* Exemestane, Letrozole, and Anastrozole belong to a class of drugs called aromatase inhibitors. the participant and the physician will choose the most appropriate aromatase inhibitor for them. These drugs act by lowering the amount of estrogen produced by the body by blocking an enzyme called aromatase. Each of these drugs have been approved by the FDA for this cancer and have been used in the treatment of metastatic ER-positive breast cancer for many years.
* In this part of the research study the investigators are looking for the safest doses of these drugs to give to participants at the same time.
* The overall goal of this study is to evaluate the safety and effectiveness of Tucatinib in combination with Abemaciclib, Trastuzumab, and hormonal therapy for hormone receptor-positive, HER2-positive Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Cohort:

* At least one measurable or non-measurable metastasis by radiographic evaluation or physical examination.
* Progressive breast cancer on most recent regimen
* Presence of CNS metastases allowed, but not required for participation in the dose escalation cohort.

Expansion Cohort A:

* At least one measurable CNS metastasis per RANO-BM, defined as ≥ 10 mm in at least one dimension.
* Unequivocal evidence of new and/or progressive brain metastases, and at least one of the following scenarios:
* Treated with SRS or surgery with residual un-treated lesions remaining. Such participants are eligible for immediate enrollment on this study providing that at least one untreated lesion is measurable
* Participants who have had prior WBRT and/or SRS and then whose lesions have subsequently progressed are also eligible. In this case, lesions which have been treated with SRS may be considered as target lesions if there is unequivocal evidence, in the opinion of the treating physician, of progression following SRS.

  * Participants who have not previously been treated with cranial radiation (e.g., WBRT or SRS) are eligible to enter the study, but such participants must be asymptomatic from their CNS metastases and not requiring corticosteroids for symptom control.
  * Both participants who present with systemic stable/absent or systemic progressive disease are eligible, as long as they fulfill one of the above criteria.

Expansion Cohort B:

* New and/or progressive brain metastasis(es) with clinical indication for surgical resection.
* Participants must have evaluable intracranial disease according to RANO-BM prior to surgical resection. Should participants also have extracranial disease, it may be evaluable according to RECIST 1.1

Expansion Cohort C:

-At least one measurable extracranial metastasis according to RECIST 1.1

All Cohorts:

* Pathologically confirmed Hormone Receptor (HR)-positive HER2-positive MBC by local laboratory with the following requirements:

  * To fulfill the requirement of HR-positive disease, the most recent biopsy (primary tumor or metastatic lesion) of the breast cancer must express at least one of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PR]) by immunohistochemistry (IHC). ER and PR assays are considered positive if there are > 1% positive tumor nuclei in the sample.
  * To fulfill the requirement of HER2-positive disease, the most recent biopsy (primary tumor or metastatic lesion) of the breast cancer must demonstrate HER2 overexpression or amplification (immunohistochemistry of 3+ or HER2 gene amplification by in situ hybridization with a ratio of HER2-gene signals to centromere 17 signals ≥ 2.0 or average HER2 copy number ≥ 6.0 signals/cells).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (echo) or multigated acquisition (MUGA) scan within 3 months before initiation of study treatment. Patients with a history of LVEF < 50% should have left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (echo) or multigated acquisition (MUGA) scan within the screening window.
* Stable or decreasing corticosteroid dose for at least 7 days prior to initiation of treatment.
* Concurrent administration of other anti-cancer therapy during the course of this study is not allowed, except for hormonal therapy with one of the commercially available aromatase inhibitors (AI) and the use of ovarian suppression in pre-menopausal patients. Note that concurrent use of supportive care medications (e.g. anti-resorptive agents, pain medications) is allowed. Pre-menopausal patients will need to receive ovarian suppression with the use of one of the commercially available GNRH agonists, per the choice of the treating physician.
* The subject is ≥18 years old.
* Participants must have normal organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1.5 × 109/L

  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 8 g/dL
* Note: Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

  * Total bilirubin ≤ 1.5 × ULN.
  * Patients with Gilbert's syndrome with a total bilirubin ≤ 2.0 times ULN and direct bilirubin within normal limits are permitted;
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 × institutional ULN.
  * Albumin > 2.5mg/dL
  * Serum creatinine ≤ 1.5 × ULN.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test prior to initiating protocol therapy.
* The effects of tucatinib, abemaciclib, and trastuzumab on the developing human fetus are unknown so women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 months after completion of tucatinib and abemaciclib administration and 7 months after trastuzumab administration.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
* Participant must be able to swallow and retain oral medication.
* Have discontinued all previous therapies for breast cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy), except for trastuzumab, for at least the following number of days prior to receiving study drug(s):

  * 28 days for myelosuppressive agents given every 28-day schedule.
  * 21 days for myelosuppressive agents given every 21-day schedule.
  * 14 days for myelosuppressive agents given every 7-day schedule, or for oral agents or for nonmyelosuppresive agents
* Patients must have recovered from the acute effects of therapy (until the toxicity resolves to either baseline or at least Grade 1) except for residual alopecia or peripheral neuropathy

Exclusion Criteria:

* Visceral crisis or impending visceral crisis at time of screening.
* CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement).
* Known leptomeningeal metastases [Defined as positive CSF cytology and/or unequivocal radiological evidence of clinically significant leptomeningeal involvement. CSF sampling is not required in the absence of suggestive symptoms to exclude leptomeningeal involvement].
* Patients unable to undergo gadolinium contrast-enhanced MRI or receive IV gadolinium contrast for any reason (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity, hypersensivity).
* Has received prior therapy with a CDK4/6 inhibitor.
* No washout is required for endocrine therapy. If a patient has been on ovarian suppression for at least 28 days prior to study entry, ccontinuation of ovarian suppression is permitted on protocol. Patients can receive a new form of endocrine therapy with one of the commercially available AIs at the time of initiation of protocol therapy.
* Subjects with a history of grade 3 or 4 allergic reactions attributed to compounds of similar biologic composition to tucatinib and/or abemaciclib or any constituent of the product(s).
* The subject has an uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, or severe malnutrition.
* The subject is pregnant or breast-feeding.1No active, second potentially life-threatening cancer. Exceptions include non-melanoma skin cancers, curatively treated in situ cancer of the cervix, DCIS, stage1/grade 1 endometrial carcinoma.
* Has had major surgery within 21 days before treatment initiation.
* Active infection requiring iv antibiotics at the time of treatment initiation.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest.
* Known intolerance to trastuzumab.
* Patients may not be receiving concurrent therapy with strong inhibitors of CYP3A4 or strong inhibitors or inducers of CYP2C8. Please refer to Appendix M for a list of inhibitors and inducers. Please note that concurrent use of trimethoprim, a component of Bactrim, is prohibited per protocol. Patients who require PCP prophylaxis will need to switch to an alternative antibiotic (e.g. mepron)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-28 (Estimated); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose | 2 years
  Determine recommended MTD for phase 2 combination of tucatinib with abemaciclib and trastuzumab.

SECONDARY OUTCOMES:
Overall Response Rate | 20 year
  Efficacy of study combination, defined by CNS ORR according to RANO-BM.
Duration of Response | 2 years
  DOR in the CNS according to RANO-BM.
Extracranial ORR | 2 Years
  Extracranial ORR according to RECIST 1.1.
Progression Free Survival | 2 years
  Bi-compartmental progression-free survival (PFS) according to RANO-BM.
Duration of Extracranial Response | 2 Years
  Duration of Extracranial Response according to RANO-BM.
Overall Survival | 2 Years
  OS will be analyzed using Kaplan-Meier product-limit estimates and 90% confidence bands
Site of First Progression | 2 Year
  Site of First Progression, CNS vs extracranial vs both
Extra-CNS response rates | 2 years
  Extra-CNS response rates according to RECIST 1.1
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  to evaluate the number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pablo Leone, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation